CLINICAL TRIAL: NCT05134649
Title: Phase 3, Multicenter Open-label Extension Study to Evaluate the Safety of BOTOX (Botulinum Toxin Type A) Purified Neurotoxin Complex for the Treatment of Platysma Prominence
Brief Title: A Study To Assess the Safety of OnabotulinumtoxinA (BOTOX) Intramuscular Injection in Adult Participants With Platysma Prominence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21-323
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Platysma Prominence
Keywords: Platysma Prominence; BOTOX; OnabotulinumtoxinA
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BOTOX (Experimental): BOTOX (OnabotulinumtoxinA) will be injected into the platysma muscle for up to 3 Cycles during study M21-323
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Intramuscular Injection
  Other Names: BOTOX

SUMMARY:
This is a Phase 3, open-label extension study to evaluate the long-term safety of repeat BOTOX treatments in adult participants with Platysma Prominence. Participants who completed the lead-in Phase 3 Study M21-309 and met eligibility requirements could enroll in this open-label extension study.

Planned study enrollment was approximately 270 participants. Participants who met treatment criteria could receive up to 3 administrations of BOTOX. Day 1 (study entry) was the same day as Day 120/study exit visit of the lead-in Phase 3 study. The first administration of study drug could occur at the Day 1 visit, and the last administration of study drug could occur at the Day 180 visit (60 days prior to Day 240/study exit). Once a subject was enrolled in this study, monthly follow-up visits occurred.

ELIGIBILITY:
Inclusion Criteria:

- Completion of all phases of the lead-in Phase 3 study (Screening Period, Treatment Period [randomization/treatment with 4-month follow-up visit] and Study Exit visit)

Exclusion Criteria:

* Any medical condition that may put the participant at increased medical risk with exposure to BOTOX, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
* Participant has an anticipated need for treatment with botulinum toxin of any serotype for any indication during the study (other than study intervention)
* Anticipated need for surgery or overnight hospitalization during the study
* Females who are pregnant or breastfeeding and are considering becoming pregnant or donating eggs during the study
* Known immunization or hypersensitivity to any botulinum toxin serotype
* History of clinically significant (per investigator's judgment) drug or alcohol abuse within the last 6 months
* Tattoos, jewelry, or clothing that cannot be removed, and that obscure the target area of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (29):
- United States (25):
  - Advanced Research Associates - Glendale /ID# 231997, Glendale, Arizona
  - Clear Dermatology & Aesthetics Center /ID# 231990, Scottsdale, Arizona
  - Clinical Testing of Beverly Hills /ID# 231986, Encino, California
  - Steve Yoelin MD Medical Assoc. Inc /ID# 232004, Newport Beach, California
  - Cosmetic Laser Dermatology /ID# 232414, San Diego, California
  - Ava T. Shamban MD - Santa Monica. /ID# 232000, Santa Monica, California
  - Art of Skin MD /ID# 231995, Solana Beach, California
  - DMR Research PLLC /ID# 231998, Westport, Connecticut
  - Susan H. Weinkle MD /ID# 232001, Bradenton, Florida
  - Research Institute of the Southeast, LLC /ID# 231974, West Palm Beach, Florida
  - Laser and Skin Surgery Center of Indiana /ID# 231983, Indianapolis, Indiana
  - Coleman Center For Cosmetic Dermatologic Surgery /ID# 231977, Metairie, Louisiana
  - Delricht Research /ID# 231985, New Orleans, Louisiana
  - Aesthetic Center at Woodholme /ID# 231996, Baltimore, Maryland
  - Maryland Dermatology Laser, Skin, & Vein Institute /ID# 232002, Hunt Valley, Maryland
  - Image Dermatology, P.C. /ID# 231980, Montclair, New Jersey
  - Laser & Skin Surgery Center of New York /ID# 231982, New York, New York
  - Aesthetic Solutions /ID# 231978, Chapel Hill, North Carolina
  - Wilmington Dermatology Center /ID# 231981, Wilmington, North Carolina
  - Aventiv Research Dublin /ID# 231994, Dublin, Ohio
  - KGL Skin Study Center, LLC /ID# 231993, Newtown Square, Pennsylvania
  - Nashville Center for Laser and Facial Surgery /ID# 231975, Nashville, Tennessee
  - Dallas Plastic Surgery Institute /ID# 231999, Dallas, Texas
  - SkinDC /ID# 231989, Arlington, Virginia
  - Premier Clinical Research /ID# 232003, Spokane, Washington
- Canada (4):
  - Humphrey Cosmetic Dermatology /ID# 239649, Vancouver, British Columbia
  - Dermetics Cosmetic Dermatology /ID# 239650, Burlington, Ontario
  - Dr Melinda Gooderham Medicine Profession /ID# 239647, Cobourg, Ontario
  - The Center For Dermatology /ID# 239651, Richmond Hill, Ontario

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 292 participants were enrolled at 28 sites in the United States and Canada. All participants received at least 1 dose of open-label BOTOX and were included in the intent-to-treat (ITT) and safety populations.
Pre-assignment Details: Safety analyses were carried out for the Safety Analysis Set (Safety Population), which consisted of all participants who received study drug in both the lead-in study and in this study (N=292).
Groups:
- BOTOX: BOTOX (OnabotulinumtoxinA) was injected into the platysma muscle for up to 3 cycles during study M21-323.
Period: Overall Study
Arm/Group | BOTOX
Started | 292
Completed | 262
Not Completed | 30
Not completed — Lost to Follow-up | 12
Not completed — Withdrawal by Subject | 14
Not completed — Pregnancy | 1
Not completed — Other, not specified | 3

BASELINE CHARACTERISTICS:
Population: ITT Population
Arm/Group | BOTOX
Number analyzed (Participants) | 292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 278
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.6 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 261
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 265
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a casual relationship with this treatment.
Time Frame: 371 days (from enrollment in the lead-in study M21-309 through end of study M21-323)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Lead-in): Participants who received placebo in M21-309 until they received their first BOTOX treatment or discontinued in M21-323.
- BOTOX (Cycle 1): Participants who received their first BOTOX treatment until they received their next BOTOX treatment or discontinued in M21-323.
  The first BOTOX treatment may have been in M21-309 or M21-323.
- BOTOX (Cycle 2): Participants who received their second BOTOX treatment until they received their next BOTOX treatment or discontinued in M21-323.
  The first BOTOX treatment may have been in M21-309 or M21-323.
- BOTOX (Cycle 3): Participants who received their third BOTOX treatment until they received their next BOTOX treatment or discontinued in M21-323.
  The first BOTOX treatment may have been in M21-309 or M21-323.
- BOTOX (Cycle 4): Participants who received their fourth BOTOX treatment until they until they discontinued or completed M21-323.
  The first BOTOX treatment was administered in M21-309.
- BOTOX (All Treatment Cycles): Participants who received at least one BOTOX treatment in either M21-309 or M21-323 and were enrolled in M21-323.
- Total: Participants who received any study drug in either M21-309 or M21-323 and were enrolled in M21-323.
Arm/Group | Placebo (Lead-in) | BOTOX (Cycle 1) | BOTOX (Cycle 2) | BOTOX (Cycle 3) | BOTOX (Cycle 4) | BOTOX (All Treatment Cycles) | Total
Number analyzed (Participants) | 151 | 292 | 268 | 177 | 54 | 292 | 292
Participants | 33 | 74 | 46 | 26 | 11 | 111 | 127

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from enrollment in M21-323 to the end of study. The median time participants were followed was 239.0 days.
Arm/Group | BOTOX
All-Cause Mortality (participants affected / at risk) | 0/292
Serious Adverse Events (participants affected / at risk) | 2/292
Other Adverse Events (participants affected / at risk) | 42/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOTOX (N=292)
CELLULITIS (Infections and infestations) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOTOX (N=292)
INJECTION SITE BRUISING (General disorders) | 12 (13)
COVID-19 (Infections and infestations) | 22 (22)
NASOPHARYNGITIS (Infections and infestations) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT05134649/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT05134649/SAP_001.pdf